CLINICAL TRIAL: NCT06490991
Title: A Clinical Study Evaluating the Relative Bioavailability of HRS-5965 Capsules and Tablets in Healthy Subjects .
Brief Title: Comparison of HRS-5965 Capsules and Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-102
Record Dates: First submitted 2024-06-23; First posted 2024-07-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria，IgA Nephropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Medication regimen 1-2 (Experimental)
  Interventions: Drug: HRS-5965 tablets；HRS-5965 capsules
- Arm B: Medication regimen 2-1 (Experimental)
  Interventions: Drug: HRS-5965 tablets；HRS-5965 capsules

INTERVENTIONS:
Drug: HRS-5965 tablets；HRS-5965 capsules — Medication regimen: 1 Drug: HRS-5965 tablets Medication regimen: 2 Drug: HRS-5965 capsules

SUMMARY:
The study is designed as a single-center, randomized, open-label, cross-over phase I clinical trial with the intention of recruiting 16 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form before the start of this trial, and be able to understand the procedures and methods of this trial. Willing to strictly follow the clinical trial protocol to complete this trial.
2. Healthy subject is male aged between 18 and 45 years (including both ends, subject to signing of informed consent form);
3. Body weight ≥ 50 kg, and body mass index (BMI): 19-26 kg/m2 (including both ends);
4. Physical examination, vital signs, 12 lead electrocardiogram, chest X-ray, abdominal ultrasound, and laboratory tests during the screening period show no abnormalities, or there are slight abnormalities that have been determined by the researcher to have no clinical significance;
5. Human immunodeficiency virus antibody (HIV Ab), treponema pallidum antibody, hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) were all negative during the screening period;
6. Male subjects with partners who are fertile women, who have no plans to conceive or donate sperm within 3 months after signing the informed consent form and voluntarily adopt efficient contraceptive measures (including partners);

Exclusion Criteria:

1. Individuals who are allergic to two or more allergens, or who have been determined by the researcher to be potentially allergic to the investigational drug or its components;
2. According to the judgment of researchers, there may be diseases or medical conditions that may affect drug absorption, distribution, metabolism, and excretion, or may reduce compliance;
3. Patients with comorbidities such as cardiovascular, liver, kidney, digestive tract, psychiatric, hematological, metabolic abnormalities, and immunodeficiency;
4. Individuals with a history of meningococcal infection or first-degree relatives with a history of meningococcal infection;
5. Screening for individuals with clear evidence of infection (positive pathogen test or previous systemic antibiotic treatment) or those with a body temperature exceeding 38 ℃ within the first two weeks;
6. Screening for individuals who have experienced severe trauma or surgery within the first 8 weeks, or plan to undergo surgery during the trial period;
7. Screening for clinical trials involving any other drugs or medical devices within the first 4 weeks or planned during the study period, or those who are still within 5 half-lives of the drugs before screening (whichever is longer);
8. Those who have used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, traditional Chinese patent medicines and simple preparations and dietary supplements) within 4 weeks before screening; Or select those who are within 5 half-lives of the drug at the time of screening (whichever is longer);
9. Those whose blood creatinine levels exceed the upper limit of normal values, or those who have not exceeded the upper limit but have been determined by the researcher to have a possibility of renal function damage;
10. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding the upper limit of normal values (ULN), or total bilirubin exceeding 1.5 times ULN;
11. When screening, individuals with QTcF>450 msec (male) , or other clinically significant abnormalities determined by the researcher;
12. Individuals with a history of blood donation or severe blood loss (blood loss ≥ 400 mL) within the 8 weeks prior to screening, or those who have received blood transfusions within the 12 weeks prior to screening;
13. Those who have used drugs or drugs in the past; Or those who tested positive for urine medication during screening;
14. Screening for individuals who smoke an average of 5 or more cigarettes per day within the first 4 weeks;
15. The average daily alcohol intake in the four weeks before screening exceeds 15 g (15 g alcohol is equivalent to 450 mL beer, 150 mL wine or 50 mL low alcohol Baijiu), or the alcohol breath test is positive during screening;
16. Difficulty swallowing, difficulty in venous blood collection, or physical condition unable to withstand blood collection; Or subjects who are expected to be unable to complete the entire trial follow-up;
17. Those who receive the vaccine within 2 weeks before the first administration or within 1 month after the last administration during the study period;
18. Subjects with a history of recurrent oral ulcers;
19. According to the judgment of the researcher, any physiological or psychological illness or condition that may increase the trial risk, affect the participant's compliance with the protocol, or affect the participant's completion of the trial, as well as any other situation determined by the researcher that the participant is not suitable to participate in the clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
The relative bioavailability (Fr) values between HRS-5965 capsules and HRS-5965 tablets taken on an empty stomach | 0-144hours
Relative bioavailability (Fr) values of HRS-5965 capsules taken on an empty stomach | 0-144hours

CONTACTS AND LOCATIONS:
Locations (1):
- ZhongShan Hospital FuDan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided